# **PROTOCOL**

**Title:** SURESTEP: Transcranial Direct Current Stimulation in Super Refractory

**Status Epilepticus (SURESTEP)** 

**Principal Investigator:** Marcus C. Ng, MD, FRCPC, CSCN; Neurology

University of Manitoba

Co-Investigators: Ji Hyun Ko, PhD; Human Anatomy and Cell Science

University of Manitoba

Bojan Paunovic, MD, FRCPC; Critical Care Medicine

University of Manitoba

NCT Number: NCT03819543

**Document Date:** February 18, 2019

## 1. Specific Aims

To investigate the efficacy of transcranial direct current stimulation (tDCS) in super refractory status epilepticus (SRSE), defined as:

- Primary Outcome #1: frequency of epileptiform activity on EEG
- Primary Outcome #2: severity of epileptiform activity on EEG (defined along the ictal-interictal continuum)

#### 2. Study Design

- i. ICU EEG Monitoring
  - The ICU team orders prolonged periods of live EEG monitoring (up to 3 hours at a time) on SRSE patients to determine:
    - whether the patient continues to seize despite the presence of ongoing intravenous anaesthetic
    - o whether it is safe to wean anaesthetic
    - o whether the patient has stopped seizing off anaesthetic
    - o if the patient has resumed seizing off anathesthic, then whether the patient is still seizing once anaesthetic is resumed.
  - During business hours, a live ICU EEG monitoring request is automatically honoured by the EEG technologist
  - After-hours (from 8 am to midnight for 7 days a week on all 365 days a year), the EEG request is first screened by the on-call neurologist
    - o If the request is approved, then the request is forwarded to the EEG technologist.

#### ii. tDCS Set-Up & Application

- tDCS will only be available when live EEG monitoring is available
  - o tDCS can only be applied maximally once a day
    - Only one tDCS session per day
    - tDCS cannot be repeated in one day
  - o tDCS can only be applied a maximum of 10 sessions over 10 days
    - Although there is no harm, there is also no perceived benefit if tDCS has not shown benefit after at least 10 sessions of stimulation
- The "HD-targets" software (Soterix Medical, New York) will be used to determine the stimulation parameters to deliver a constant current of 2.0 mA at the epileptogenic foci for 20 minutes
  - HD-targets uses a model human brain to estimate the focal delivery of direct current by adjusting current intensity of 8 channels.
  - If the epileptogenic focus is diffuse or cannot be identified from EEG, then tDCS shall be applied to the right (nondominant) temporal pole

### iii. Real-Time Anaesthetic Management

- Once the EEG technologist has finished their typical clinical set-up, live EEG data will start streaming to a non-blinded EEG reader (an epileptologist or a neurologist with special interest in EEG) at a remote location for interpretation.
- Based on the EEG reader's live report(s) to the ICU team, anaesthetic(s) may be changed
  - o If the ICU elects to make no anaesthetic changes, then tDCS shall be applied right away
  - o If the ICU elects to increase or decrease anaesthetic, then another 10 minutes shall elapse for the anaesthetic change to take effect prior to tDCS application
- During real-time tDCS application, the EEG reader will determine efficacy by assessing whether there has been enough improvement in the frequency and severity of epileptiform activity (primary study outcomes #1 and #2) to warrant discontinuation (or continued discontinuation) of intravenous anaesthetic sedation to the end of the EEG recording (secondary study outcome)
  - Frequency of epileptiform activity (primary outcome #1) is defined as the number of discharges per unit time (e.g. spikes per minute)
  - Severity of epileptiform activity (primary outcome #2) is defined by the morphology of the activity as outlined by the American Clinical Neurophysiology Society Standardized Critical Care EEG Terminology for the interictal-ictal continuum (e.g. spikes or sharp waves are more epileptiform than broad sharp waves or sharply contoured activity)
  - o If tDCS unexpectedly worsens epileptiform activity, tDCS will be terminated immediately
- After tDCS application is complete, the RA will remove all tDCS equipment from the patient and the bedside
- The EEG reader will continue live-monitoring the study to ensure that any changes in the frequency and/or severity of epileptiform activity are enduring (i.e. persist through to the end of EEG recording)
- Total EEG recording will be 3 hours as per the usual maximum ICU EEG recording duration protocol

#### 3. Statistical Analysis Plan

- The primary study outcomes of epileptiform activity frequency before, during, and after tDCS will be analyzed on a per-stimulation session basis
- The primary study outcomes of epileptiform activity frequency before, during, and after tDCS will also be analyzed on a per-patient session basis by averaging spike rates for all sessions in that patient
- All data will be assessed for normality using the Shapiro-Wilk test

• Parametric tests will be used for normally distributed data and non-parametric tests will be used for non-normally distributed data in order to test before vs. during tDCS on persession and per-patient bases; and before vs. after tDCS on per-session and per-patient bases